CLINICAL TRIAL: NCT05996458
Title: A Population-based, Multicenter Cohort Study of Combined Screening for Gastrointestinal Tumors
Status: Recruiting | Type: Observational
Sponsor: Xijing Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: KY20232111-F-1号
Record Dates: First submitted 2023-08-10; First posted 2023-08-18 (Actual); Last update posted 2023-10-11 (Actual); Status verified 2023-07

CONDITIONS: Digestive Disease
MeSH Terms: conditions — Digestive System Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood；tissue
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- group one: The screening population will undergo gastroscopy, colonoscopy, fecal occult blood test (FIT), Helicobacter pylori (HP) antigen test, ring finger protein 180 (RNF180) and SEPTIN9 gene methylation test, and investigation of risk factors, including past disease history, alcohol drinking history, smoking history, tea drinking history, family history of cancer, marital and reproductive status, and dietary habits.
  Interventions: Other: Gastroenteroscopy；Risk factor investigation; FIT-HP;RNF180 and SEPTIN9 gene methylation test
- Group one's control（Spouse or sibling of group one ): Only the risk factors will be investigated
  Interventions: Other: Risk factor investigation;
- group two: The screening population will undergo investigation of risk factors, a fecal occult blood test (FIT), and a stool test for Helicobacter pylori (HP) antigen. If a stool occult blood test or H. pylori antigen is positive after testing, RNF180 and SEPTIN9 gene methylation testing will be scheduled. If the gene methylation test is positive, a colonoscopy will be scheduled.
  Interventions: Other: Gastroenteroscopy；Risk factor investigation; FIT-HP;RNF180 and SEPTIN9 gene methylation test
- group two's control（Spouse or sibling of group two): Only the risk factors will be investigated
  Interventions: Other: Risk factor investigation;

INTERVENTIONS:
Other: Gastroenteroscopy；Risk factor investigation; FIT-HP;RNF180 and SEPTIN9 gene methylation test — group one: The screening population will undergo gastroscopy, colonoscopy, fecal occult blood test (FIT), Helicobacter pylori (HP) antigen test, RNF180/Septin9 gene methylation test, and investigation of risk factors, including past disease history, alcohol drinking history, smoking history, tea drinking history, family history of cancer, marital and reproductive status, and dietary habits.
  Groups: group one
Other: Risk factor investigation; — Only the risk factors will be investigated, including previous disease history, drinking history, smoking history, drinking history, family history of malignant tumor, marriage and childbearing status, eating habits, etc.
  Groups: Group one's control（Spouse or sibling of group one ); group two's control（Spouse or sibling of group two)
Other: Gastroenteroscopy；Risk factor investigation; FIT-HP;RNF180 and SEPTIN9 gene methylation test — group two: The screening population will undergo investigation of risk factors, a fecal occult blood test (FIT), and a stool test for Helicobacter pylori (HP) antigen. If a stool occult blood test or H. pylori antigen is positive after testing, RNF180 and SEPTIN9 gene methylation testing will be scheduled. If the gene methylation test is positive, a colonoscopy will be scheduled.
  Groups: group two

SUMMARY:
To establish combined gastroenteroscopy screening and follow-up management for gastrointestinal tumors, explore and evaluate the feasibility and health economic benefits of combined screening for esophagus, stomach and colorectal cancer

DETAILED DESCRIPTION:
group one: The screening population will undergo gastroscopy, colonoscopy, fecal occult blood test (FIT), Helicobacter pylori (HP) antigen test, ring finger protein 180 (RNF180) and SEPTIN9 gene methylation test, and investigation of risk factors, including past disease history, alcohol drinking history, smoking history, tea drinking history, family history of cancer, marital and reproductive status, and dietary habits.

group two: The screening population will undergo investigation of risk factors, a fecal occult blood test (FIT), and a stool test for Helicobacter pylori (HP) antigen. If a stool occult blood test or H. pylori antigen is positive after testing, RNF180 and SEPTIN9 gene methylation testing will be scheduled. If the gene methylation test is positive, a colonoscopy will be scheduled.

Group one's control（Spouse or sibling of group one);group two's control（Spouse or sibling of group one): Only the risk factors will be investigated, including previous disease history, drinking history, smoking history, drinking history, family history of malignant tumor, marriage and childbearing status, eating habits, etc.

Finally, 10 years follow-up will be conducted to observe the outcome

ELIGIBILITY:
Inclusion Criteria:

* 1. Subjects were 45 to 70 years old when enrolled 2. Willing and able to sign informed consent

Exclusion Criteria:

* 1. History of any type of malignancy 2. Previous resection of esophagus, stomach or colorectal 3. Received gastrointestinal endoscopy such as colonoscopy and gastroscopy in recent 5 years 4. Have received fecal occult blood test and fecal DNA test in the past 1 year. 5. Contraindications to endoscopy. 6. Warning symptoms of digestive tract tumors, including:

  1. Difficulty swallowing, choking or halting feeling when eating recently
  2. Recent esophageal foreign body sensation or swallowing pain
  3. Recent long-term loss of appetite and appetite
  4. Recent and prolonged symptoms of indigestion (including acid reflux, heartburn, abdominal grumbling, burping, nausea or premature satiety, etc.)
  5. Recent symptoms of abdominal mass, abdominal pain, vomiting or hematemesis
  6. It was medically diagnosed as iron deficiency anemia
  7. Recent changes in hematochezia, black stool or stool character and frequency
  8. Recent symptoms of perianal discomfort (including soreness, itching, lumps, prolapse or other discomfort)
  9. Unexplained weight loss (more than 10% of base body weight) in the past 6 months Step 7 Get pregnant 8. There are other serious comorbiditions that reduce screening benefits (including severe lung disease, advanced kidney disease, advanced liver disease, severe heart failure, etc.)

Ages: 45 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Eligible Chinese persons
Sampling Method: Probability Sample
Enrollment: 84000 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2032-11-30 (Estimated); Study Completion 2033-06-30 (Estimated)

PRIMARY OUTCOMES:
Cancer or precancerous lesions detected | 10 year
  Cancer or precancerous lesions detected

CONTACTS AND LOCATIONS:
Overall Officials: Kaichun Wu, Study Chair — Xijing Hospital
Locations (1):
- Gaoyao District People's Hospital, Zhaoqing, Guangzhou, China

IPD SHARING:
Plan to Share IPD: Undecided
According to the research process, choose a specific method to disclose the original data.